CLINICAL TRIAL: NCT06430723
Title: Obesity and it's Impact on Subsidence and Clinical Outcomes After Short Stem Total Hip
Brief Title: The Impact of Obesity on Short Stem Total Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: Krankenhaus Barmherzige Schwestern Linz (Other)
Responsible Party: Sponsor
Other Study IDs: EK 1258/2023
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: THA; Obesity
Keywords: subsidence; obesity; short stem total hip arthroplasty; tha
MeSH Terms: conditions — Obesity | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-obese: Body mass index < 30 kg/m2
  Interventions: Procedure: Total hip arthroplasty
- Obese: Body mass index >= 30 kg/m2
  Interventions: Procedure: Total hip arthroplasty

INTERVENTIONS:
Procedure: Total hip arthroplasty — Total hip arthroplasty using short stem via an minimally invasive anterolateral approach

SUMMARY:
The purpose of this study is to review the impact of obesity on subsidence and clinical outcome after short stem total hip arthroplasty.

DETAILED DESCRIPTION:
Short stem total hip arthroplasty (THA) has gained popularity due to its bone-sparing technique, but its outcomes in obese patients remain uncertain.

While studies on the mid-term outcome in a general patient cohort provide excellent results in terms of the clinical and radiological outcome as well as the complication rate of short stem THA, data on its use in obese patients is still rare and not sufficiently conclusive. Some studies have found no evidence of increased subsidence in obese patients, while other studies have shown contrary trends.

In this context, the aim of this study was to investigate the relationship between BMI, postoperative subsidence and clinical outcomes in the setting of short stem THA.

ELIGIBILITY:
Inclusion Criteria:

1. patients who underwent primary short stem hip arthroplasty with Mathys Optimys short stem between 01.01.2018 and 31.12.2020
2. availability of preoperative and postoperative radiographs for assessment of subsidence
3. a minimum BMI of 30kg/m2 for the obese group
4. a minimum follow-up of 24 months.

Exclusion Criteria:

1. former surgeries of the hip in question
2. incomplete clinical data
3. incomplete radiological data

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The purpose of this study was to assess the subsidence rates in patients who underwent short stem hip arthroplasty and its association with obesity. To investigate this, an analysis of patient data was conducted together with a follow-up examination, focusing on clinical outcome and radiographic analysis of the subsidence of the stem in obese patients. Hence, two groups based on body mass index were retrospectively evaluated: obese (BMI ≥ 30 kg/m^2) and non-obese (BMI < 30 kg/m^2), with an age of minimum 18 years, but no maximum age.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Subsidence | 2 years
  subsidence of the short stem measured via EBRA (Einzelbild Röntgenanalyse), [mm]
Harris Hip Score | 2 years
  Clinical outcome, [0-100points]

SECONDARY OUTCOMES:
surgery time | 2 years
  Surgery time from cut to skin closure, [minutes]
Length of stay | 2 years
  Length of postoperative stay in hospital [days]
Blood loss | 2 years
  Blood loss calculated according to laboratory test results of hematocrit [ml]

CONTACTS AND LOCATIONS:
Locations (1):
- Ordensklinikum Linz, Barmherzige Schwestern Abteilung Orthopädie, Linz, Austria

IPD SHARING:
Plan to Share IPD: No